CLINICAL TRIAL: NCT01858493
Title: Phase 3 Cluster Randomised Trial Testing the Efficacy of a Continence Promotion Intervention to Improve Urinary Symptoms and Quality of Life, and Reduce Stigma and Falls in Older Community-dwelling Women With Untreated Incontinence
Brief Title: Continence Across Continents to Upend Stigma and Dependency
Acronym: CACTUS-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government); Medical Research Council (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government); Institut national de prevention et d'education pour la sante (Other Government)
Responsible Party: Principal Investigator, Cara Tannenbaum, Principal Investigator, Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ERA-AGE2 dossier28835
Record Dates: First submitted 2013-05-14; First posted 2013-05-21 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Urinary Incontinence; Falls, Accidental; Quality of Life; Stigma
Keywords: Urinary incontinence; Falls; Quality of life; Stigma; Community-dwelling older women; Continence promotion
MeSH Terms: conditions — Urinary Incontinence; Social Stigma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continence promotion group education (Experimental): A single 1-hour continence promotion group education workshop, facilitated by the research coordinator, aimed at changing knowledge and beliefs about urinary incontinence and different treatment options. An evidence-based self-management tool will be distributed at the end of the workshop.
  Interventions: Behavioral: Continence promotion group education workshop
- Sham health lecture (Sham Comparator): A single 1-hour group education workshop on other health topics of concern to older women such as memory, hearing, insomnia
  Interventions: Behavioral: Sham health lecture

INTERVENTIONS:
Behavioral: Continence promotion group education workshop — Interactive group education workshop promoting continence
  Arms: Continence promotion group education
Behavioral: Sham health lecture — Interactive group education workshop about general health
  Arms: Sham health lecture

SUMMARY:
To determine whether women exposed to the continence promotion intervention will report improved urinary symptoms and quality of life, and lower incontinence-related stigma and falls than women who receive a control intervention at one-year post-intervention.

DETAILED DESCRIPTION:
This is a cluster-randomized 4-site intervention study testing the effect of a continence-promotion intervention on:

1. Improved urinary symptoms and quality of life
2. Reduction in falls
3. Reduction in stigma

A cost-effectiveness component will also be included

ELIGIBILITY:
Inclusion Criteria:

* Women
* 65 years and older
* Urinary incontinence at least once weekly

Exclusion Criteria:

* Living in residential or long-term care
* Received treatment for incontinence within the past year
* Dementia or other neurological conditions that preclude the ability to provide -Informed consent

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 910 (Actual)
Dates: Start 2013-05; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Self-reported improvement in urinary incontinence | 1 year
  Patient global impression of improvement questionnaire Sandvik severity index ICIQ-FLUTS

SECONDARY OUTCOMES:
Falls | 1 year
  Reduction in incontinence-related falls measured by fall diary
Reduction in incontinence related stigma and quality of life | 1 year
  Measured with the Incontinence Quality of Life questionnaire (IQOL)

OTHER OUTCOMES:
Cost-utility of the continence promotion intervention | 1-year
  Cost/QALY. Direct costs will include costs related to the intervention as well as health care resource use due to incontinence-associated falls and health care seeking for incontinence will be measured. Indirect costs will be measured such as the time lost from work for a child or spouse to accompany the participant to receive medical treatment for incontinence or falls. The change in utility from the baseline incontinent condition to improved incontinence with increased social participation and decreased stigma on quality of life will be calculated from SF6D utilities derived from the SF-12 questionnaire at baseline and 1-year follow-up. A disease-specific measure, the IQOL is currently undergoing mapping onto the SF-6D to see if it will provide a more responsive indication of improved quality of life than the generic SF-12 measure.

CONTACTS AND LOCATIONS:
Overall Officials: Cara Tannenbaum, MD. MSc, Principal Investigator — Univeristé de Montréal; Adrian Wagg, MD, Principal Investigator — University of Alberta; Eleanor van den Heuvel, PhD, Principal Investigator — Brunel University; Xavier Fritel, MD, PhD, Principal Investigator — University of Poitiers
Locations (4):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Institut universitaire de gériatrie de Montréal, Montreal, Quebec
- Université de Poitiers, Poitiers, Poitou-Charentes, France
- University of Brunel, Uxbridge, Middlesex, United Kingdom

REFERENCES:
- [Background] Agnew R, van den Heuvel E, Tannenbaum C. Efficiency of using community organisations as catalysts for recruitment to continence promotion trials. Clin Trials. 2013 Feb;10(1):151-9. doi: 10.1177/1740774512460144. Epub 2012 Oct 5. PMID 23043154
- [Background] Tannenbaum C, Agnew R, Benedetti A, Thomas D, van den Heuvel E. Effectiveness of continence promotion for older women via community organisations: a cluster randomised trial. BMJ Open. 2013 Dec 10;3(12):e004135. doi: 10.1136/bmjopen-2013-004135. PMID 24334159
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568
- [Derived] Tannenbaum C, van den Heuvel E, Fritel X, Southall K, Jutai J, Rajabali S, Wagg A. Continence Across Continents To Upend Stigma and Dependency (CACTUS-D): study protocol for a cluster randomized controlled trial. Trials. 2015 Dec 10;16:565. doi: 10.1186/s13063-015-1099-x. PMID 26652168